CLINICAL TRIAL: NCT06910722
Title: Liver Transplantation for Locally Advanced Intrahepatic Cholangiocarcinoma After Selective Internal Radiotherapy With Labeled Yttrium and Chemotherapy: a Phase 2 Study
Brief Title: Liver Transplantation for Locally Advanced Intrahepatic Cholangiocarcinoma After SIRT and Chemotherapy
Acronym: RIS-TH
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: APHP220677
Record Dates: First submitted 2025-03-28; First posted 2025-04-04 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-03

CONDITIONS: Liver Transplantation in Locally Advanced Intrahepatic Cholangiocarcinoma
Keywords: liver transplantation; locally advanced intrahepatic cholangiocarcinoma; selective internal radiation therapy
MeSH Terms: interventions — Liver Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- liver transplant patients (Experimental): Liver transplantation performed after selective internal radiotherapy (SIRT) with Yttrium-90 and chemotherapy in patients with locally advanced (unresectable but non-metastatic) intrahepatic cholangiocarcinoma.
  Interventions: Procedure: Liver transplant

INTERVENTIONS:
Procedure: Liver transplant — follow-up of liver transplant patients after selective internal radiotherapy (SIRT) with Yttrium-90 and chemotherapy

SUMMARY:
The study hypothesis is that liver transplantation after selective internal radiation therapy (SIRT) and chemotherapy would improve 3-year overall survival in patients with locally advanced (unresectable but non-metastatic) intrahepatic cholangiocarcinoma.

It is planned to include 36 patients with locally advanced intrahepatic cholangiocarcinoma, not eligible for initial surgery and without metastases. Participants will be recruited from care facilities in France.

DETAILED DESCRIPTION:
The hypothesis of the study is that liver transplantation after selective internal radiation therapy (SIRT) and chemotherapy would improve the overall 3-year survival of patients with locally advanced intrahepatic cholangiocarcinoma (unresectable but not metastatic).

All patients over 18 and under 65 years of age with histologically evidence, pauci-nodular (N≤5), locally advanced Intrahepatic cholangiocarcinoma (IHC) without extrahepatic involvement, considered technically unresectable by a panel of experts, eligible for treatment with SIRT, gemcitabine + cisplatin chemotherapy and Liver Transplant (LT).

Following treatment with SIRT + chemotherapy, tumor response or absence of tumor progression will be verified by a morphological workup combining CT-imaging, hepatic MRI and PET-CT.

After exploratory surgery to rule out any contraindications for LT, the patient will be list , with a minimum waiting of 3-month Follow-up will include assesment of Liver graft function, efficiency and tolerance of immunosuppressive therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 to 65
* With histologically documented intrahepatic cholangiocarcinoma (primary diagnosis):

  * Uni or pauci nodular (≤ 5 lesions (all lesions are counted, even those less than 1 cm))
  * Without extrahepatic or lymph node involvement
  * Technically unresectable R0 according to an expert panel
* Tumor target > 2 cm
* WHO 0-1
* free and informed consent signed
* highly effective contraception for men and women of childbearing age during study participation up to 2 years post TH

Exclusion Criteria:

* Extrahepatic, vesicular or perihilar cholangiocarcinoma
* Tumor infiltration of more than 50% of the liver
* Mixed cholangiocarcinoma, hepatocellular carcinoma, fibrolamellar carcinoma
* Previous treatment for CCI
* Cirrhosis ≥ Child B7
* Chronic alcoholism
* Uncontrolled chronic active infections (patients with HBV, HCV or HDV infections may be included if infections are controlled)
* Stage III A, IIIB, IV and V chronic renal failure (glomerular filtration rate 59 ml/min)
* Contraindications to liver transplant

  * Severe untreatable conditions
  * Recent history (less than 5 years) of cancer
  * severe comorbidities
  * Psychiatric or psychological disorders
* Pregnant or breast-feeding women
* Patient under guardianship
* Not affiliated to a Health care system
* Participating in another interventional study or within the exclusion period of a previous study involving the human body

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2028-04-01 (Estimated); Study Completion 2030-04-01 (Estimated)

PRIMARY OUTCOMES:
Strategy efficacy : 3 years overall survival | 3 years post-transplant
  To assess the 3-year overall survival of patients undergoing liver transplantation for stable or downstaged locally advanced intrahepatic cholangiocarcinoma after induction treatment with selective internal radiotherapy and chemotherapy.

SECONDARY OUTCOMES:
Strategy feasibility 1/2 | Liver transplantation
  Number of patients benefiting from the complete strategy implemented
Strategy feasibility 2/2 contraindication to transplantation | Liver transplantation
  Number of patients with radiological tumor progression according to RECIST 1.1 criteria after neoadjuvant treatment contraindicating transplantation
Associated factors with the 3-years overall survival | 3 years after strategy implementation
  Socio-demographic and clinico-radio-biological characteristics at baseline and follow-up of living patients 3 years after strategy implementation.
therapeutic efficacy at 3 years | 3 years after strategy implementation
  Number of transplant patients alive and free of recurrence at 3 years after strategy implementation, as well as their socio-demographic and clinico-radiobiological characteristics at baseline and follow-up.
therapeutic efficacy at 5 years | 5 years after strategy implementation
  Number of transplanted patients alive 5 years after the strategy was implemented and number of transplanted patients alive and free of recurrence for the same period;.
oncological prognosis1/2 | after 8 courses of chemotherapy
  Number of patients not transplanted alive at 3 years (with or without recurrence)
oncological prognosis 2/2 | 5 years after strategy implementation
  Time to onset, type and location of recurrence in transplanted and non-transplanted patients
Histological response | 1 year after strategy implementation
  Rate of tumor necrosis on total hepatectomy specimens in transplant patients
Tolerance of neoadjuvant treatment | after 8 courses of chemotherapy
  Number and type of adverse events induced by neoadjuvant therapy
quality of life monitoring | from induction therapy until 5 years post-transplant
  Changes in scores on the SF-36 quality-of-life questionnaire administered after neoadjuvant treatment prior to TH and then annually between the first and fifth years of follow-up
Tolerance of global strategy | from induction therapy until 3 months post-transplant
  Number of adverse events of grade greater than or equal to 3 (NCI CTCAE) during neoadjuvant treatment + Number of severe complications greater than or equal to 3 of the Clavien-Dindo classification within 90 days of TH.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Bouattour, Principal Investigator — APHP